CLINICAL TRIAL: NCT02078076
Title: IRM Cardiaque en Respiration Libre Pour Des Patients Atteints de Dystrophinopathie sévère
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C13-04; 2013-A00179-36 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-06-03; First posted 2014-03-05 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2016-02

CONDITIONS: Duchenne or Severe Becker Myopathy
Keywords: MRI; free-breathing acquisitions; myopathy; fibrosis assessment; function
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Diseases; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic Resonance Cardiac Imaging (with Gadolinium) (Experimental)
  Interventions: Device: Magnetic Resonance Cardiac Imaging (with Gadolinium)

INTERVENTIONS:
Device: Magnetic Resonance Cardiac Imaging (with Gadolinium)

SUMMARY:
Clinical, prospective and monocentric study aiming at assessing the feasibility of fibrosis detection and quantification (and of function assessment) during MRI without breath-holds in a population of adults and children with Duchenne myopathy.

ELIGIBILITY:
Inclusion Criteria:

* Dystophinopathy (Duchenne or severe Becker)
* >8yo
* with social insurance
* informed consent

Exclusion Criteria:

* arythmia
* impossibility to undergo an MRI (pacemaker, ....)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of exams correctly acquired (feasabiliy of the exam) | after the last inclusion
  Was it possible to acquire the whole examination for every patient ?
Number of exams allowing a qualitative assessment of images by the physician | after the last MRI exam
  The image quality allows a qualitative diagnosis ?
Number of exams allowing a quantitative assessment of the diagnosis | after the last MRI examination
  Did the image quality allow a quantitative assessment of the diagnosis ?

SECONDARY OUTCOMES:
Number of anatomic cardiac segments with significant fibrosis according to the assessment methods (conventional LGE, qualitative detection with GRICS, and quantiative measure with GRICS) | after the last inclusion
  correlation between fibrosis information (conventional LGE, qualitative detection with GRICS, and quantiative measure with GRICS)
Number of cardiac segments with fibrosis and/or regional dysfunction | after the last inclusion
  Correlation between fibrosis and regional function for each cardiac segment

CONTACTS AND LOCATIONS:
Locations (1):
- Service de médecin nucléaire / CHU Nancy Brabois, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Background] Odille F, Bustin A, Liu S, Chen B, Vuissoz PA, Felblinger J, Bonnemains L. Isotropic 3D cardiac cine MRI allows efficient sparse segmentation strategies based on 3D surface reconstruction. Magn Reson Med. 2018 May;79(5):2665-2675. doi: 10.1002/mrm.26923. Epub 2017 Oct 2. PMID 28971520